CLINICAL TRIAL: NCT07360782
Title: Individualized Application of Occipital Nerve Pulsed Radiofrequency in Medication Overuse Headache: A Randomized Controlled Evaluation
Brief Title: Personalized Pulsed Radiofrequency of the Greater Occipital Nerve for Medication Overuse Headache
Acronym: PRIMOGON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Şükriye Dadalı, Pain Medicine (Algology) specialist, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2-25-12241
Record Dates: First submitted 2026-01-10; First posted 2026-01-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Medication Overuse Headache
Keywords: Medication Overuse Headache; Occipital Nerve Pulsed Radiofrequency; Headache Treatment
MeSH Terms: conditions — Headache Disorders, Secondary | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants are initially randomized in a parallel design to receive either standard treatment alone or standard treatment plus greater occipital nerve pulsed radiofrequency (GONPRF). An adaptive second stage is applied at the 1-month assessment, in which participants who do not respond adequately to standard treatment receive GONPRF as a second-line intervention, while follow-up continues in parallel groups.
Masking Description: This is an open-label study. No participants, care providers, investigators, or outcome assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1- Standard Treatment (Group A1) (Experimental): Intervention Name: Standard Care Intervention Type: Other (Behavioral / Educational / Non-drug) Description: Limitation of overused acute headache medications, lifestyle advice (nutrition, hydration, activity, sleep), and continuation of preventive medications. Participants who respond at 1 month continue standard care.
  Interventions: Other: Standard care
- Arm 2: Primary GONPRF (Group B) (Experimental): Intervention Name: Greater Occipital Nerve Pulsed Radiofrequency (GONPRF)
  Intervention Type: Procedure
  Description: GONPRF applied at C2 under ultrasound guidance in addition to standard care, starting at enrollment. Follow-up at 1, 3, and 6 months.
  Interventions: Procedure: Greater Occipital Nerve Pulsed Radiofrequency
- Arm 3: Modified GONPRF (Group A2) (Experimental): Intervention Name: Greater Occipital Nerve Pulsed Radiofrequency (GONPRF) - Second Line
  Intervention Type: Procedure
  Description: Participants initially on standard care who do not achieve ≥50% improvement at 1 month receive GONPRF as a second-line intervention, alongside continued standard care, with follow-up at 3 and 6 months.
  Interventions: Procedure: Greater Occipital Nerve Pulsed Radiofrequency

INTERVENTIONS:
Procedure: Greater Occipital Nerve Pulsed Radiofrequency — GONPRF applied at C2 under ultrasound guidance in addition to standard care, starting at enrollment. Follow-up at 1, 3, and 6 months.
  Arms: Arm 2: Primary GONPRF (Group B); Arm 3: Modified GONPRF (Group A2)
Other: Standard care — Limitation of overused acute headache medications, lifestyle advice (nutrition, hydration, activity, sleep), and continuation of preventive medications. Participants who respond at 1 month continue standard care.
  Arms: Arm 1- Standard Treatment (Group A1)

SUMMARY:
This study evaluates a novel treatment approach for medication overuse headache (MOH) using greater occipital nerve pulsed radiofrequency (GONPRF).

Three treatment strategies are compared:

Standard Treatment: Limitation of overused acute headache medications, lifestyle counseling, and continuation of existing preventive medications.

Primary GONPRF: GONPRF administered in addition to standard treatment.

Modified GONPRF: GONPRF administered as a second-line intervention in individuals who do not respond adequately to standard treatment alone.

The study assesses whether GONPRF, when applied early or after an initial period of standard care, reduces monthly headache days more rapidly and effectively than standard treatment alone. Outcomes are evaluated over a 6-month follow-up period using headache diaries and scheduled clinical assessments.

This is a randomized controlled trial designed to systematically evaluate the clinical benefit of GONPRF in patients with medication overuse headache.

DETAILED DESCRIPTION:
This is a single-center, prospective, adaptive randomized controlled trial evaluating the efficacy of greater occipital nerve pulsed radiofrequency (GONPRF) in patients with medication overuse headache (MOH). Although occipital nerve blocks have been investigated in MOH, randomized controlled trials evaluating GONPRF in this population are lacking. The study aims to compare different treatment strategies incorporating GONPRF in the management of MOH.

Study Design

The trial employs a two-stage adaptive randomized design.

Stage 1 - Initial Randomization

Patients diagnosed with MOH according to the International Classification of Headache Disorders, 3rd edition (ICHD-3), are randomized in a 2:1 ratio into two groups:

Standard Treatment Group: Limitation of overused acute headache medications, lifestyle recommendations (including nutrition, hydration, physical activity, and sleep hygiene), and continuation of ongoing preventive medications without dose modification.

Primary GONPRF Group: Ultrasound-guided GONPRF applied at the C2 level in addition to standard treatment.

Stage 2 - One-Month Assessment

At one month, all patients are evaluated for predefined primary and secondary outcome measures, including monthly headache days, headache intensity, number of days requiring acute medication, Headache Impact Test (HIT-6), and Global Perceived Effect (GPE) scores.

Patients in the Standard Treatment Group who fail to achieve a ≥50% improvement in at least one primary outcome measure receive GONPRF as a second-line intervention and are classified as the Modified GONPRF Group. Patients demonstrating adequate response continue standard treatment and are classified as Standard Treatment Responders.

Patients initially randomized to the Primary GONPRF Group continue follow-up without additional intervention modifications.

Follow-Up and Data Collection

All interventions are performed on an outpatient basis. Follow-up assessments are conducted at baseline and at 1, 3, and 6 months. Patients maintain daily headache diaries documenting headache occurrence, intensity, duration, and use of acute headache medications. Diary data are supplemented by structured clinical evaluations at each follow-up visit.

Adaptive Outcome Classification

Following the one-month assessment, patients are categorized into three groups:

Standard Treatment Responders (Group A1)

Modified GONPRF Group (Group A2)

Primary GONPRF Group (Group B)

The final distribution among the three groups is anticipated to be approximately equal.

Acute Medication Protocol

Patients receive structured counseling regarding limitation of overused acute headache medications. Alternative short-acting analgesic or antimigraine medications may be used, limited to a maximum of two days per week. Preventive medications in use at baseline are continued without dose adjustment throughout the study period.

Study Purpose

The primary objective is to evaluate the clinical efficacy of GONPRF in the treatment of medication overuse headache when applied either as an early adjunctive therapy or as a second-line intervention following standard care. A secondary objective is to assess whether the timing of GONPRF initiation influences clinical outcomes.

ELIGIBILITY:
Inclusion Criteria

* Age 18-65 years
* Diagnosed with Medication Overuse Headache (MOH) according to ICHD-3 criteria
* No laboratory evidence of bleeding or clotting disorders
* No active infection
* Not pregnant and no suspicion of pregnancy
* No history of craniocervical surgery that may alter anatomical structures at the intervention site
* Able to understand the study procedures, provide written informed consent, and comply with treatment

Exclusion Criteria

* Changes in preventive treatment for migraine and/or tension-type headache within the last 3 months
* Severe systemic disease (e.g., uncontrolled diabetes, serious cardiovascular disease, malignancy)
* Psychiatric disorders (including current antidepressant use or psychiatric follow-up)
* History of alcohol or substance abuse
* Pregnancy, breastfeeding, or plans for pregnancy in the next 12 months
* Concurrent use of other prophylactic headache treatments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Monthly Headache Days | Baseline to 3 months
  Number of headache days per month, defined as days with headache lasting ≥4 hours and/or requiring acute headache treatment, recorded using patient headache diaries. The primary analysis compares the change from baseline to 3 months.

SECONDARY OUTCOMES:
Monthly Headache Days - 1 and 6 Months | Baseline, 1 month, and 6 months
  Number of headache days per month assessed at early and longer-term follow-up time points to evaluate short- and long-term treatment effects.
Monthly Acute Medication Use Days | Baseline, 1 month, 3 months, and 6 months
  Number of days per month on which acute headache medications (paracetamol, nonsteroidal anti-inflammatory drugs, triptans, ergot derivatives, or opioids) are used, as recorded in headache diaries.
Headache Pain Intensity (Numeric Rating Scale, NRS) | Baseline, 1 month, 3 months, and 6 months
  Average and maximum headache pain intensity per attack measured using the 11-point Numeric Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst possible pain. Higher scores represent greater pain severity.
Headache Duration (hours) | Baseline, 1 month, 3 months, and 6 months
  Average duration of each headache attack in hours.
Headache Impact Test-6 (HIT-6) Score | Baseline, 1 month, 3 months, and 6 months
  Headache Impact Test-6 (HIT-6) total score, range 0-78, measuring the impact of headaches on daily activities, social functioning, work, and quality of life. Higher scores indicate greater headache-related disability (worse outcome).
Migraine Disability Assessment (MIDAS) Grade | Baseline, 3 months, and 6 months
  Migraine Disability Assessment (MIDAS) evaluates headache-related disability over the past 3 months. Scores are categorized into four grades:
  Grade I: Minimal or infrequent disability Grade II: Mild disability Grade III: Moderate disability Grade IV: Severe disability Higher grades indicate greater disability (worse outcome). Participants will be assessed at baseline, 3 months, and 6 months.
Global Perceived Effect (GPE) Score | Baseline, 1 month, 3 months, and 6 months
  Global Perceived Effect (GPE) is a 7-point Likert scale measuring overall change in the patient's main complaint and general well-being. Scores range from 1 (much worse) to 7 (much improved), with higher scores indicating greater improvement.

OTHER OUTCOMES:
GONPRF Treatment Side (Unilateral/Bilateral) | During the GONPRF procedure (Day 1 of intervention)
  Side of the greater occipital nerve treated during the pulsed radiofrequency procedure, recorded as left, right, or bilateral.
Adverse Events Related to GONPRF | From the time of the GONPRF procedure through study completion (up to 6 months).
  All procedure-related adverse events (e.g., injection site pain, infection, vasovagal reaction) will be recorded, including type, severity, and duration.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not planned due to national regulations regarding patient data confidentiality.

REFERENCES:
- [Background] Gosalia H, Moreno-Ajona D, Goadsby PJ. Medication-overuse headache: a narrative review. J Headache Pain. 2024 May 31;25(1):89. doi: 10.1186/s10194-024-01755-w. PMID 38816828
- [Background] Ashina S, Terwindt GM, Steiner TJ, Lee MJ, Porreca F, Tassorelli C, Schwedt TJ, Jensen RH, Diener HC, Lipton RB. Medication overuse headache. Nat Rev Dis Primers. 2023 Feb 2;9(1):5. doi: 10.1038/s41572-022-00415-0. PMID 36732518